CLINICAL TRIAL: NCT06245382
Title: The Impact of Goode Health Beverage on Markers of Physiological and Neurocognitive
Brief Title: The Impact of Goode Health Beverage on Markers of Physiological and Neurocognitive Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Matthew Brothers, Professor, The University of Texas at Arlington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-0202
Record Dates: First submitted 2024-01-29; First posted 2024-02-07 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases; Hypertension; Cognitive Decline; Diet, Healthy
Keywords: endothelial function, brain blood flow, cognition
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Individuals will be randomly assigned to either an experimental or a control condition.
Who Masked: Investigator
Masking Description: This will be a double-blinded design where the product (experimental of control) will be randomly assigned and given to the participant by a third party individual.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Goode Health Beverage (Experimental): Goode Health Beverage that is high in natural ingredients that are high in Polyphenol 3 content and also have anti-inflammatory and antioxidant properties
  Interventions: Dietary Supplement: Goode Health Beverage
- Vanilla Base Blend Beverage (Placebo Comparator): The control beverage is similar but it does not contain the same amount of fiber, anti-inflammatory, and/or antioxidant properties (i.e. mainly smaller or no amounts of flax, ginger, cinnamon, turmeric, berberine bergamot, bilberry, black garlic, and green tea).
  Interventions: Dietary Supplement: Vanilla Base Beverage Blend

INTERVENTIONS:
Dietary Supplement: Goode Health Beverage — This is a commercially available beverage powder that is high is healthy ingredients that are believed to be beneficial for physiological health.
  Arms: Goode Health Beverage
Dietary Supplement: Vanilla Base Beverage Blend — This is a commercially available beverage powder.
  Arms: Vanilla Base Blend Beverage

SUMMARY:
The overall research objective of this proposal is to determine the acute and chronic impact of daily supplementation of a Good Health beverage on indices of physiological and neurocognitive health.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of morbidity and mortality and affects all individuals. There are many primary risk factors for CVD with some of the primary causes including hypertension, hypercholesteremia, atherosclerosis, and type 2 diabetes mellitus. Furthermore, the rise in the prevalence of various neurocognitive conditions and cerebral vascular diseases including cognitive dysfunction, dementia, stroke, and Alzheimer's disease requires additional attention from a research perspective. While the reasons contributing to CVD and neurocognitive complications/cerebral vascular diseases, is multifactorial, a common link is impaired vascular function.

A hallmark of impaired vascular function is elevated arterial stiffness and a decrease in the vasodilator capacity in the brain and periphery. Reduced nitric oxide (NO) bioavailability, due to elevated oxidative stress and systemic inflammation is implicated as a primary contributing factor for these attenuated vasodilatory responses. Therefore, it is reasonable to speculate that an approach targeting these pathways could abolish or minimize this elevated risk. One such approach could be increased dietary consumption of a naturally based product that is high in polyphenol content and ingredients that are well-known to have beneficial effects on oxidative stress, inflammation, blood lipids etc. In turn this would be expected to have beneficial outcomes on various biomarkers associated with peripheral and cerebral vascular health including, cholesterol, lipid profile, insulin sensitivity/type II diabetes, cognitive health, arterial stiffness, blood pressure, and NO bioavailability and subsequently vascular function/health. Specifically, the Goode Health Super Food Smoothie Blend is a product that we are interested in investigating in this proposal.

1. Primary Aim - The primary endpoint is the effect of increased daily consumption of the Good Health beverage on outcomes associated with elevated risk for various neurocognitive and pathophysiological conditions/diseases. These outcomes include cognitive function, central and peripheral arterial blood pressure, cerebral and peripheral blood vessel function/health, and blood biomarkers (e.g., indices of inflammation, oxidative stress, insulin resistance/diabetes risk, and lipid profile).
2. Secondary Aim - A secondary endpoint is the effect of daily consumption of the Good Health beverage on the following variables: waist circumference, body weight, and body mass index (BMI).

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are between the ages of 18-55

Exclusion Criteria:

* Individuals who have donated more than 550 ml of blood within the past 8 weeks will not have blood drawn from them in this protocol. However, if they remain interested in the study, and otherwise meet the inclusion criteria, then we may still opt to proceed with data collection.
* Any food allergy.
* Pregnant women
* Breast feeding
* Allergies to spandex/lycra.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Endothelial Function | baseline & following 2 weeks of daily beverage consumption
  Flow medicated dilation of the brachial artery
Neurocognitive Function | baseline & following 2 weeks of daily beverage consumption
  Performance on the NIH Toolbox Cognitive battery
Peripheral blood pressure (systolic, diastolic, mean) | baseline & following 2 weeks of daily beverage consumption
  standard blood pressure measures
Lipid profile (Total-C, LDL-C, VLDL-C, HDL-C, TG) | baseline & following 2 weeks of daily beverage consumption
  assessment of lipid profile

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Brothers, PhD, Principal Investigator — University of Texas at Arlington
Locations (2):
- United States (2):
  - UT Arlington - Science and Engineering Innovation and Research Building, Arlington, Texas
  - UT Arlington, Arlington, Texas

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IDP.